CLINICAL TRIAL: NCT05414643
Title: Management of Acute Cardiogenic Shock at the New Brunswick Heart Centre
Acronym: Team-Shock
Status: Completed | Type: Observational
Sponsor: New Brunswick Heart Centre (Other)
Responsible Party: Principal Investigator, Dr. Jean-François Légaré, Head of Cardiac Surgery, New Brunswick Heart Centre
Other Study IDs: 101097
Record Dates: First submitted 2022-04-14; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Cardiogenic Shock
Keywords: mortality; outcomes; AMI; shock team; SCAI stage; intervention; IABP; ECMO
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- At- risk group (SCAI stages A, B): Patients who had a SCAI stage A or B at any point during their stay at the New Brunswick Heart Centre, Saint John Regional Hospital. This group was compared with the cardiogenic shock group only for preliminary analysis.
  Interventions: Other: Standard care
- Cardiogenic shock group (SCAI stages C-E): Patients who had a SCAI (Society for Cardiovascular Angiography and Interventions) stage C-E at any point during their stay at the New Brunswick Heart Centre, Saint John Regional Hospital. This group was used for all subsequent analyses.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — No interventions were used, as this is an observational study.

SUMMARY:
In Atlantic Canada, acute myocardial infarction occurs at a rate of 2.9 % of the population and is the most common cause of cardiogenic shock (CS). In many studies, acute myocardial infarction accounts for up to 80% of the patients with CS. While there are different methods of treating patients with CS, the rate of mortality has not significantly improved over the years and remains as high as 50%. Recent studies have shown that a multi-modal, team-based approach can help improve patient outcomes; however, such a standardized approach is yet to be implemented in the New Brunswick Heart Centre (NBHC).

The study aims to understand the difference in outcomes between two groups of patients treated for CS: SHOCK TEAM versus non-SHOCK TEAM. This is a retrospective study of 168 patients using the data from NBHC registry and patient charts. The study duration is 1 year. The primary outcome is hospital survival. Secondary outcomes include time from diagnosis to invasive monitoring and intervention. All data will be analyzed statistically between the two groups. The end goal of the study is to establish standard guidelines to treat CS patients and improve patient survival.

ELIGIBILITY:
Inclusion Criteria:

1) Any patient admitted to the CCU with a diagnosis of CS (SCAI groups C, D or E) at any point during their CCU care.

Exclusion Criteria:

1) CS patients having SCAI groups A, B (this group was used only for preliminary analysis, hence this is the exclusion criteria for all final analyses).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who were admitted to the CCU at the NBHC, Saint John Regional Hospital between November 1st 2019 to November 30th 2020 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1416 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Percentage mortality | From the date of hospital admission at Saint John Regional Hospital to the date of discharge, assessed upto 6 months
  Any in-hospital mortality (within Saint John Regional Hospital, another hospital after transfer)
Length of stay (LOS)) | From the date of hospital admission at Saint John Regional Hospital to the date of discharge, assessed upto 6 months
  LOS was considered only for patients who were discharged directly home from Saint John Regional Hospital
Discharge disposition | From the date of hospital admission at Saint John Regional Hospital to the date of discharge, assessed upto 6 months
  Discharge of patients home, transfer to another hospital or to another institution (special care home, extra-mural home)
Percentage of missed opportunities | From the date of hospital admission at Saint John Regional Hospital to the date of discharge, assessed upto 6 months
  Missed opportunities was defined as patients who suffered significant delays or those who did not receive any intervention

SECONDARY OUTCOMES:
Time from diagnosis of shock to in-hospital processes | From the date of hospital admission at Saint John Regional Hospital to the date of discharge, assessed upto 6 months
  Time gaps between the first diagnosis of a cardiogenic shock to in-hospital processes like invasive monitoring, cardiac catheterization or interventions (surgery, PCI, TAVI, IABP or ECMO).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Légaré, M.D., Ph.D., Principal Investigator — New Brunswick Heart Centre
Locations (1):
- New Brunswick Heart Centre, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No